CLINICAL TRIAL: NCT02333071
Title: Phase 3, Randomized, Double-blind, Placebo-controlled, Trial With an Open-label Extension Phase to Evaluate the Efficacy and Safety of Subcutaneously Bremelanotide in Premenopausal Women With Hypoactive Sexual Desire Disorder (HSDD)
Brief Title: 1. Study to Evaluate the Efficacy/Safety of Bremelanotide in Premenopausal Women With Hypoactive Sexual Desire Disorder
Acronym: HSDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Palatin Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMT-301; Reconnect Study (Other: Palatin Technologies, Inc.)
Record Dates: First submitted 2014-12-28; First posted 2015-01-07 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2020-12

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: HSDD; Female Sexual Desire Disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — bremelanotide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bremelanotide (BMT/BMT) (Experimental): (Main Study) Subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 24 weeks
  (OLE Study) Subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 52 weeks
  Interventions: Drug: Bremelanotide
- Placebo (PBO/BMT) (Placebo Comparator): (Main Study) PBO administered SC on an as-desired basis for 24 weeks
  (OLE Study) subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 52 weeks
  Interventions: Drug: Bremelanotide; Other: Placebo

INTERVENTIONS:
Drug: Bremelanotide — A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
  Other Names: BMT; PT-141
Other: Placebo — Placebo
  Other Names: PBO
  Arms: Placebo (PBO/BMT)

SUMMARY:
A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial with an optional Open-label Extension to evaluate the efficacy of bremelanotide (BMT), administered subcutaneously (SC) on an as needed basis for the treatment of HSDD (with or without decreased arousal) in premenopausal females.

DETAILED DESCRIPTION:
This will be a multicenter, randomized, placebo-controlled, parallel group study in up to 80 sites in the United States of America (USA) and Canada to evaluate the efficacy and safety of a fixed dose of SC BMT versus placebo on an as-needed basis under conditions of home use in premenopausal women with HSDD (with or without decreased arousal).

The study will consist of 2 phases: (1) Core Study: 4-week no-treatment qualification period, a 4-week single-blind placebo treatment period (baseline), and a 24-week double-blind treatment period where participants will self-administer placebo or BMT 1.75 mg SC via an autoinjector; and (2) Extension Phase: a 52-week open-label treatment period during which all subjects will receive BMT 1.75 mg.

Primary Objective

• To evaluate the efficacy of bremelanotide (BMT), administered subcutaneously (SC) on an as needed basis for the treatment of HSDD (with or without decreased arousal) in premenopausal females.

Secondary Objectives

* To evaluate the efficacy of BMT in premenopausal women in the double-blind Core Study, as assessed by subject responses to questionnaires measuring sexual function, treatment satisfaction, and distress associated with sexual dysfunction.
* To evaluate the safety of BMT in premenopausal women in the double-blind Core Study.
* To evaluate the safety of long-term therapy with BMT in the open label Extension Phase.
* To evaluate the efficacy of long-term therapy with BMT in the open-label Extension Phase.

ELIGIBILITY:
Main Inclusion Criteria:

* Has met diagnostic criteria for HSDD for at least 6 months
* Is willing and able to understand and comply with all study requirements
* Has a normal pelvic examination at screening

Main Exclusion Criteria:

* Subjects should be generally healthy premenopausal females with no psychological, gynecological or urological conditions which might contribute to the sexual dysfunction, compromise study participation, or confound interpretation of the study results
* Not currently under treatment for the sexual dysfunction and willing to forego other treatments through the course of the clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 723 (Actual)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jordan, Study Director — Palatin Technologies, Inc
Locations (91):
- United States (87):
  - Palatin Clinical Site 121, Birmingham, Alabama
  - Palatin Clinical Site 110, Huntsville, Alabama
  - Palatin Clinical Site 106, Mobile, Alabama
  - Palatin Clinical Site 149, Scottsdale, Arizona
  - Palatin Clinical Site 157, Tucson, Arizona
  - Palatin Clinical Site 166, Little Rock, Arkansas
  - Palatin Clinical Site 102, National City, California
  - Palatin Clinical Site 164, Oceanside, California
  - Palatin Clinical Site 152, Orange, California
  - Palatin Clinical Site 188, Sacramento, California
  - Palatin Clinical Site 141, San Diego, California
  - Palatin Clinical Site 187, Walnut Creek, California
  - Palatin Clinical Site 160, Centennial, Colorado
  - Palatin Clinical Site 185, Colorado Springs, Colorado
  - Palatin Clinical Site 130, Bradenton, Florida
  - Palatin Clinical Site 128, Hollywood, Florida
  - Palatin Clinical Site 134, Jacksonville, Florida
  - Palatin Clinical Site 108, Melbourne, Florida
  - Palatin Clinical Site 105, Orlando, Florida
  - Palatin Clinical Site 131, South Miami, Florida
  - Palatin Clinical Site 144, St. Petersburg, Florida
  - Palatin Clinical Site 101, West Palm Beach, Florida
  - Palatin Clinical Site 116, Decatur, Georgia
  - Palatin Clinical Site 142, Savannah, Georgia
  - Palatin Clinical Site 171, Meridian, Idaho
  - Palatin Clinical Site 179, Evansville, Indiana
  - Palatin Clinical Site 165, Lafayette, Indiana
  - Palatin Clinical Site 154, Mishawaka, Indiana
  - Palatin Clinical Site 184, West Des Moines, Iowa
  - Palatin Clinical Site 155, Overland Park, Kansas
  - Palatin Clinical Site 104, Wichita, Kansas
  - Palatin Clinical Site 191, Louisville, Kentucky
  - Palatin Clinical Site 194, Eunice, Louisiana
  - Palatin Clinical Site 186, New Orleans, Louisiana
  - Palatin Clinical Site 183, Bangor, Maine
  - Palatin Clinical Site 159, Annapolis, Maryland
  - Palatin Clinical Site 119, Boston, Massachusetts
  - Palatin Clinical Site 126, Watertown, Massachusetts
  - Palatin Clinical Site 163, Bingham Farms, Michigan
  - Palatin Clinical Site 181, Rochester, Michigan
  - Palatin Clinical Site 182, Olive Branch, Mississippi
  - Palatin Clinical Site 170, St Louis, Missouri
  - Palatin Clinical Site 180, Billings, Montana
  - Palatin Clinical Site 192, Norfolk, Nebraska
  - Palatin Clinical Site 168, Omaha, Nebraska
  - Palatin Clinical Site 111, Las Vegas, Nevada
  - Palatin Clinical Site 125, Las Vegas, Nevada
  - Palatin Clinical Site 109, Las Vegas, Nevada
  - Palatin Clinical Site 195, Las Vegas, Nevada
  - Palatin Clinical Site 120, Moorestown, New Jersey
  - Palatin Clinical Site 123, Plainsboro, New Jersey
  - Palatin Clinical Site 124, Albuquerque, New Mexico
  - Palatin Clinical Site 189, Johnson City, New York
  - Palatin Clinical Site 107, New York, New York
  - Palatin Clinical Site 158, Port Jefferson, New York
  - Palatin Clinical Site 127, Poughkeepsie, New York
  - Palatin Clinical Site 190, Rochester, New York
  - Palatin Clinical Site 137, Charlotte, North Carolina
  - Palatin Clinical Site 135, Winston-Salem, North Carolina
  - Palatin Clinical Site 156, Winston-Salem, North Carolina
  - Palatin Clinical Site 139, Fargo, North Dakota
  - Palatin Clinical Site 140, Akron, Ohio
  - Palatin Clinical Site 122, Beachwood, Ohio
  - Palatin Clinical Site 151, Cincinnati, Ohio
  - Palatin Clinical Site 112, Columbus, Ohio
  - Palatin Clinical Site 115, Englewood, Ohio
  - Palatin Clinical Site 132, Medford, Oregon
  - Palatin Clinical Site 146, Portland, Oregon
  - Palatin Clinical Site 169, Jenkintown, Pennsylvania
  - Palatin Clinical Site 172, Media, Pennsylvania
  - Palatin Clinical Site 117, Warwick, Rhode Island
  - Palatin Clinical Site 162, Anderson, South Carolina
  - Palatin Clinical Site 143, Bluffton, South Carolina
  - Palatin Clinical Site 114, Mt. Pleasant, South Carolina
  - Palatin Clinical Site 145, Mt. Pleasant, South Carolina
  - Palatin Clinical Site 161, Memphis, Tennessee
  - Palatin Clinical Site 129, Nashville, Tennessee
  - Palatin Clinical Site 174, Bryan, Texas
  - Palatin Clinical Site 113, Dallas, Texas
  - Palatin Clinical Site 118, San Antonio, Texas
  - Palatin Clinical Site 176, Sugar Land, Texas
  - Palatin Clinical Site 100, Murray, Utah
  - Palatin Clinical Site 103, Charlottesville, Virginia
  - Palatin Clinical Site 138, Virginia Beach, Virginia
  - Palatin Clinical Site 133, Spokane, Washington
  - Palatin Clinical Site 150, Tacoma, Washington
  - Palatin Clinical Site 193, Middleton, Wisconsin
- Canada (4):
  - Palatin Clinical Site 304, Halifax, Nova Scotia
  - Palatin Clinical Site 303, Kentville, Nova Scotia
  - Palatin Clinical Site 301, Toronto, Ontario
  - Palatin Clinical Site 302, Saint Romuald, Quebec

REFERENCES:
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Derived] Spielmans GI, Ellefson EM. Small Effects, Questionable Outcomes: Bremelanotide for Hypoactive Sexual Desire Disorder. J Sex Res. 2024 May;61(4):540-561. doi: 10.1080/00224499.2023.2175192. Epub 2023 Feb 21. PMID 36809187
- [Derived] Clayton AH, Kingsberg SA, Portman D, Sadiq A, Krop J, Jordan R, Lucas J, Simon JA. Safety Profile of Bremelanotide Across the Clinical Development Program. J Womens Health (Larchmt). 2022 Feb;31(2):171-182. doi: 10.1089/jwh.2021.0191. PMID 35147466
- [Derived] Koochaki P, Revicki D, Wilson H, Pokrzywinski R, Jordan R, Lucas J, Williams LA, Sadiq A, Krop J. The Patient Experience of Premenopausal Women Treated with Bremelanotide for Hypoactive Sexual Desire Disorder: RECONNECT Exit Study Results. J Womens Health (Larchmt). 2021 Apr;30(4):587-595. doi: 10.1089/jwh.2020.8460. Epub 2021 Feb 3. PMID 33538638
- [Derived] Revicki DA, Althof SE, Derogatis LR, Kingsberg SA, Wilson H, Sadiq A, Krop J, Jordan R, Lucas J. Reliability and validity of the elements of desire questionnaire in premenopausal women with hypoactive sexual desire disorder. J Patient Rep Outcomes. 2020 Oct 8;4(1):82. doi: 10.1186/s41687-020-00241-6. PMID 33033885
- [Derived] Simon JA, Kingsberg SA, Portman D, Williams LA, Krop J, Jordan R, Lucas J, Clayton AH. Long-Term Safety and Efficacy of Bremelanotide for Hypoactive Sexual Desire Disorder. Obstet Gynecol. 2019 Nov;134(5):909-917. doi: 10.1097/AOG.0000000000003514. PMID 31599847
- [Derived] Kingsberg SA, Clayton AH, Portman D, Williams LA, Krop J, Jordan R, Lucas J, Simon JA. Bremelanotide for the Treatment of Hypoactive Sexual Desire Disorder: Two Randomized Phase 3 Trials. Obstet Gynecol. 2019 Nov;134(5):899-908. doi: 10.1097/AOG.0000000000003500. PMID 31599840
- [Derived] Clayton AH, Lucas J, DeRogatis LR, Jordan R. Phase I Randomized Placebo-controlled, Double-blind Study of the Safety and Tolerability of Bremelanotide Coadministered With Ethanol in Healthy Male and Female Participants. Clin Ther. 2017 Mar;39(3):514-526.e14. doi: 10.1016/j.clinthera.2017.01.018. Epub 2017 Feb 9. PMID 28189361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Core ("Main") Study consisted of a 4-week no drug Screening period, followed by a 4-week single blind PBO period, first dose administered in-clinic. Following the end of single-blind period, which served as Baseline, eligible subjects were then randomized to a 24-week double-blind outpatient treatment period, first dose administered in-clinic.
Pre-assignment Details: Core Study: 723 participants enrolled, 70 run-in failures 653 participants were randomized.
  OLE Study (optional): Of the 464 completers of the Core study, 363 participants enrolled in optional OLE study. The OLE study was not reported and has no NCT number.
Groups:
- Placebo PBO/BMT: Core Study: Subjects will self-administer a fixed dose of placebo subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 24 weeks.
  Placebo
  OLE Study: Subjects will self-administer a fixed dose of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 52 weeks.
  bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
- Bremelanotide BMT/BMT: Core and OLE Study: Subjects will self-administer a fixed dose of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 24 weeks.
  bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
Period: Core Study
Arm/Group | Placebo PBO/BMT | Bremelanotide BMT/BMT
Started | 326 | 327
Received Intervention | 319 | 324
Completed | 274 | 190
Not Completed | 52 | 137
Period: Open Label Extension
Arm/Group | Placebo PBO/BMT | Bremelanotide BMT/BMT
Started (363/464 subjects who completed Core Study continued to this OLE Study (124 BMT-BMT and 239 PBO-BMT. The OLE study was not reported.) | 239 | 124
Completed | 95 | 49
Not Completed | 144 | 75

BASELINE CHARACTERISTICS:
Population: A total of 653 subjects were randomized into the double-blind period of the study; 10 subjects were not dosed, therefore total = 643. A total of 363 of the 464 (78.2%) subjects who completed the Core Study Phase continued into the optional OLE Study Phase.
Groups:
- Bremelanotide (BMT/BMT): Subjects will self-administer a fixed dose of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours (Main) followed by a 52-week open label extension study (OLE)
  BMT/BMT
  bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
- Placebo (PBO/BMT): Subjects will self-administer a fixed dose of placebo (PBO) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours (Main) followed by a 52-week open label extension study (OLE) where participants receive only BMT, no placebo
  PBO/BMT
  Placebo: Placebo bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
- Total: Total of all reporting groups
Arm/Group | Bremelanotide (BMT/BMT) | Placebo (PBO/BMT) | Total
Number analyzed (Participants) | 324 | 319 | 643
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: A total of 363 of the 464 subjects who completed the Core Study Phase continued into the optional OLE Study Phase, including 124 in the BMT (BMT/BMT) group and 239 in the PBO (PBO/BMT) group.
  Years
    Main | 38.4 (6.95) | 38.5 (7.22) | 38.5 (7.08)
    OLE: number analyzed (Participants) | 124 | 239 | 363
    OLE | 38.5 (6.72) | 38.8 (6.93) | 38.7 (6.85)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A total of 363 of the 464 subjects who completed the Core Study Phase continued into the optional OLE Study Phase, including 124 in the BMT (BMT/BMT) group and 239 in the PBO (PBO/BMT) group.
  Participants
    Main: Female | 324 | 319 | 643
    Main: Male | 0 | 0 | 0
    OLE: number analyzed (Participants) | 124 | 239 | 363
    OLE: Female | 124 | 239 | 363
    OLE: Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 363 of the 464 subjects who completed the Core Study Phase continued into the optional OLE Study Phase, including 124 in the BMT (BMT/BMT) group and 239 in the PBO (PBO/BMT) group.
  Participants
    Main: Hispanic or Latino | 33 | 31 | 64
    Main: Not Hispanic or Latino | 291 | 288 | 579
    Main: Unknown or Not Reported | 0 | 0 | 0
    OLE: number analyzed (Participants) | 124 | 239 | 363
    OLE: Hispanic or Latino | 13 | 20 | 33
    OLE: Not Hispanic or Latino | 111 | 219 | 330
    OLE: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 363 of the 464 subjects who completed the Core Study Phase continued into the optional OLE Study Phase, including 124 in the BMT group and 239 in the PBO group
  Participants
    Main: American Indian or Alaska Native | 3 | 1 | 4
    Main: Asian | 2 | 3 | 5
    Main: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Main: Black or African American | 44 | 42 | 86
    Main: White | 273 | 269 | 542
    Main: More than one race | 1 | 3 | 4
    Main: Unknown or Not Reported | 1 | 1 | 2
    OLE: number analyzed (Participants) | 124 | 239 | 363
    OLE: American Indian or Alaska Native | 2 | 0 | 2
    OLE: Asian | 2 | 2 | 4
    OLE: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    OLE: Black or African American | 17 | 29 | 46
    OLE: White | 101 | 204 | 305
    OLE: More than one race | 1 | 3 | 4
    OLE: Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of a Fixed Dose of Bremelanotide as Measured by FSFI (Question Q1 and Q2), 28-day Recall.
Description: As measured by change from baseline to end-of-study in the desire domain from the FSFI (Question Q1 and Q2), 28-day recall, co-primary endpoint - FSFI desire domain.
  FSFI = Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. Its six subscales assess desire, arousal, lubrication, orgasm, satisfaction, and pain, by summing individual items that comprise the subscale and multiplying the sum by a factor, resulting in a score ranging from 1.2 to 6. Increasing scores on this scale represent an increase in sexual desire and is a positive outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: A total of 363 of the 464 subjects who completed the Core Study Phase continued into the optional OLE Study Phase, including 124 in the BMT/BMT group and 239 in the PBO/BMT group.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Bremelanotide BMT/BMT: (Main Study) Subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 24 weeks
  (OLE Study) Subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 52 weeks
  bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
- Placebo PBO/BMT: (Main Study) PBO administered SC on an as-desired basis for 24 weeks
  Placebo: Placebo
  (OLE Study) subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 52 weeks
  Bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 313 | 315
score on a scale
  Main study | 0.54 (1.106) | 0.24 (0.994)
  Open label extension: number analyzed (Participants) | 49 | 97
  Open label extension | 1.30 (1.105) | 0.77 (1.138)

2. Primary Outcome: Efficacy of a Fixed Dose of Bremelanotide as Measured by FSDS-DAO (Item 13)
Description: As measured by the change from baseline to End-of-Study of the Core Study in the bothered by low desire item from the FSDS-DAO (Female Sexual Distress Scale - Desire Arousal Orgasm) (item 13).: co-primary endpoint - FSDS-DAO bothered by low desire item 13.
  Responses range from 0 (never) to 4 (always). Decreasing scores on this scale represent an increase in sexual desire (positive outcome).
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: A total of 363 of the 464 (78.2%) subjects who completed the Core Study Phase continued into the optional OLE Study Phase.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 313 | 314
score on a scale
  Main study | -0.73 (1.203) | -0.36 (1.082)
  Open label extension: number analyzed (Participants) | 49 | 97
  Open label extension | -1.7 (1.21) | -0.9 (1.10)

3. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by the Change in Baseline to End of Study in the Number of Satisfying Sexual Events (SSEs) Associated With Study Drug Administration
Description: Patient's change, from baseline to end of study (EOS), in the number of Satisfying Sexual Events (SSEs), as measured by a response of 'Yes' to question 10 (Q10) of the Female Sexual Encounter Profile-Revised questionnaire (FSEP-R). The end point was calculated as the number of events during the last 4 weeks of treatment with Q10 = Yes minus the number of baseline events with Q10 = Yes.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: A total of 363 of the 464 (78.2%) subjects who completed the Core Study Phase continued into the optional OLE Study Phase. 146 participants in the OLE study completed the 52 weeks.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 314 | 316
events
  Main study | 0.0 (1.44) | -0.1 (1.35)
  Open label extension: number analyzed (Participants) | 49 | 97
  Open label extension | 0.28 (1.457) | 0.10 (1.189)

4. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by a Change From Baseline to End of Study in Mean Desire Score (Q3) From FSEP-R
Description: Scores range from 0 (no desire) to 3 (high desire) for an individual encounter. Change from baseline is computed as the mean of the scores from all encounters for a subject in the last 28 days minus the mean of the scores from all encounters for the subject in the last 28 days before Visit 3. Only FSEP-R data pertaining to encounters recorded within 72 hours of the encounter are included.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 314 | 316
score on a scale
  Main study | 0.0 (1.09) | 0.1 (0.92)
  Open label extension: number analyzed (Participants) | 49 | 97
  Open label extension | 0.66 (0.975) | 0.38 (1.107)

5. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by a Change From Baseline to End of Study in Mean Satisfaction With Desire Score (Q4) From FSEP-R
Description: Patient's change, from baseline to end of study (EOS), in mean satisfaction with desire score, as measured by a response to question 4 (Q4) of the Female Sexual Encounter Profile-Revised questionnaire (FSEP-R). Responses range from 1 (Not at all satisfied) to 4 (Completely satisfied).
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 314 | 316
score on a scale
  Main study | 0.2 (1.15) | 0.0 (0.96)
  Open label extension: number analyzed (Participants) | 49 | 97
  Open label extension | 0.93 (1.141) | 0.59 (1.054)

6. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by a Change From Baseline to End of Study in the FSDS-DAO Total Score
Description: FSDS-DAO = Female Sexual Distress Scale - Desire/Arousal/Orgasm Scores range from 0 (never feel bothered) to 60 (always feel bothered).
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 313 | 314
score on a scale
  Main study | -9.2 (13.86) | -5.5 (12.27)
  Open label extension: number analyzed (Participants) | 49 | 97
  Open label extension | -21.4 (13.96) | -12.0 (13.66)

7. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by a Change From Baseline to End of Study in the Total FSFI Total Score
Description: FSFI = Female Sexual Function Index: a multidimensional self-report instrument for the assessment of female sexual function.
  The FSFI total score is on a scale ranging from 2 to 36. Increasing scores on this scale represent an increase in sexual desire and is a positive outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 313 | 315
score on a scale
  Main study | 2.69 (7.317) | 0.95 (5.963)
  Open label extension: number analyzed (Participants) | 49 | 97
  Open label extension | 7.71 (8.076) | 3.95 (6.740)

8. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by a Change From Baseline to End of Study in the Mean Level of Sexual Arousal (Q6) From the FSEP-R
Description: FSEP-R=Female Sexual Encounter Profile - Revised Scores range from 0 (not at all aroused) to 3 (highly aroused) for an individual encounter. A higher score indicates a better outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 314 | 316
score on a scale
  Main study | 0.1 (1.11) | -0.1 (0.93)
  Open label extension: number analyzed (Participants) | 49 | 97
  Open label extension | 0.65 (1.035) | 0.43 (1.029)

9. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by a Change From Baseline to End of Study in the Mean Satisfaction With Sexual Arousal (Q7) From the FSEP-R
Description: as for outcome 8
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 314 | 316
score on a scale
  Main study | 0.2 (1.20) | -0.1 (1.02)
  Open label extension: number analyzed (Participants) | 49 | 97
  Open label extension | 0.99 (1.170) | 0.60 (1.116)

10. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by a Change From Baseline to End of Study in the Scored Time Spent Being Concerned by Difficulty With Sexual Arousal (Q14) From the FSDS-DAO
Description: FSDS-DAO = Female Sexual Distress Scale-Desire/Arousal/Orgasm. The outcome reported is the mean score from the 15-item self assessment. The result is on a scale ranging from 0 ("never") to 4 ("always").
  A higher score indicates a worse outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 313 | 314
score on a scale
  Main study | -0.6 (1.24) | -0.4 (1.07)
  Open label extension: number analyzed (Participants) | 49 | 97
  Open label extension | -1.5 (1.23) | -1.0 (1.12)

11. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by a Change From Baseline to End of Study in the Arousal Domain of the FSFI (Q3 to Q6)
Description: FSFI = Female Sexual Function Index: a multidimensional self-report instrument for the assessment of female sexual function.
  The score is on a scale ranging from 1.2 to 6. Increasing scores on this scale represent an increase in sexual desire and is a better outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 313 | 315
score on a scale
  Main study | 0.66 (1.596) | 0.16 (1.240)
  Open label extension: number analyzed (Participants) | 49 | 97
  Open label extension | 1.46 (1.724) | 1.08 (1.581)

12. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by a Change From Baseline to End of Study in the Total Number of SSEs
Description: Change from Baseline to EOS in the total number of satisfying sexual events SSEs that occurred within 16 hours of a study drug dosing and reported within 72 hours. A higher value indicates a better outcome.
Time Frame: 8 weeks baseline plus 24 weeks (Main Study), 52 Weeks (OLE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Bremelanotide BMT/BMT | Placebo PBO/BMT
Number analyzed (Participants) | 314 | 316
events
  Main study | -0.1 (1.76) | -0.2 (1.79)
  Open label extension: number analyzed (Participants) | 49 | 97
  Open label extension | 0.65 (1.676) | 0.05 (1.553)

13. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by a Change From Baseline to End of Study in the Desire Domain of the FSFI (Q1 to Q2) Throughout the Entirety of the Double-blind Phase
Description: FSFI = Female Sexual Function Index: a multidimensional self-report instrument for the assessment of female sexual function.
  The score is on a scale ranging from 1.2 to 6. Increasing scores on this scale represent an increase in sexual desire and is a positive outcome.
Time Frame: 24 weeks (Main Study)
Population: Number of participants in just the double-blind study. The OLE study was not a double-blind study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Bremelanotide BMT: (Main Study) Subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 24 weeks
  bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
- Placebo PBO: (Main Study) PBO administered SC on an as-desired basis for 24 weeks
  Placebo: Placebo
Arm/Group | Bremelanotide BMT | Placebo PBO
Number analyzed (Participants) | 192 | 272
score on a scale | 0.69 (1.114) | 0.23 (0.933)

14. Secondary Outcome: Change From Baseline to End of Study in the Total Score for FSDS-DAO (Item 13) Throughout the Entirety of the Double-blind Phase
Description: FSDS-DAO = Female Sexual Distress Scale - Desire/Arousal/Orgasm. The FSDS-DAO is a validated 15-item self-assessment of sexual feelings and problems. The score is on a scale ranging from 0 ("never") to 4 ("always"). A higher score indicates a worse outcome.
  The score is the mean change from Baseline observed at EOS (Baseline score - EOS score) for FSDS-DAO Item 13 (feeling bothered by low sexual desire).
Time Frame: 24 weeks (Main Study)
Population: Number of participants in just the double-blind study. The OLE study was not a double-blind study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo PBO: Subjects will self-administer a fixed dose of placebo subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours.
  Placebo: Placebo
Arm/Group | Bremelanotide BMT | Placebo PBO
Number analyzed (Participants) | 192 | 271
score on a scale | -0.9 (1.23) | -0.3 (1.05)

15. Secondary Outcome: Efficacy of a Fixed Dose of Bremelanotide, as Measured by a Change From Baseline to End of Study in the Number of SSEs Associated With Study Drug Administration Throughout the Entirety of the Double-blind Phase
Description: Mean change from Baseline to EOS in the number of satisfying sexual events SSEs that occurred within 16 hours of study drug dosing and reported within 72 hours. An increase in number reflects a positive outcome.
Time Frame: 24 weeks (Main Study)
Population: Number of participants in just the double-blind study. The OLE study was not a double-blind study.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Bremelanotide BMT | Placebo PBO
Number analyzed (Participants) | 193 | 276
events | 0.1 (1.66) | -0.1 (1.37)

ADVERSE EVENTS:
Time Frame: 6 months (Main study), 12 months (Open Label study)
Description: Reporting participants: all subjects who were randomized and used at least 1 dose of double-blind study drug.
Groups:
- Bremelanotide (Main Study): Subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 24 weeks.
  bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
- Placebo (Main Study): Subjects will self-administer a fixed dose of placebo subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours.
  Placebo: Placebo
- Bremelanotide (OLE): Subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours for 52 weeks
  bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
- Placebo (OLE): Subjects will self-administer a fixed dose of bremelanotide (BMT) subcutaneously (SC) via auto-injector on an as needed basis with no more than 1 dose taken every 24 hours f or 52 weeks.
  bremelanotide: A melanocortin agonist and synthetic peptide analog of the naturally occurring hormone alpha-MSH (melanocyte-stimulating hormone)
Arm/Group | Bremelanotide (Main Study) | Placebo (Main Study) | Bremelanotide (OLE) | Placebo (OLE)
All-Cause Mortality (participants affected / at risk) | 0/324 | 0/319 | 0/124 | 0/239
Serious Adverse Events (participants affected / at risk) | 4/324 | 1/319 | 0/124 | 2/239
Other Adverse Events (participants affected / at risk) | 255/324 | 160/319 | 95/124 | 200/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bremelanotide (Main Study) (N=324) | Placebo (Main Study) (N=319) | Bremelanotide (OLE) (N=124) | Placebo (OLE) (N=239)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritoneal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometriosis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bremelanotide (Main Study) (N=324) | Placebo (Main Study) (N=319) | Bremelanotide (OLE) (N=124) | Placebo (OLE) (N=239)
Flushing (Vascular disorders) | 84 | 2 | 24 | 65
Headache (Nervous system disorders) | 32 | 8 | 13 | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 2 | 9
Nausea (Gastrointestinal disorders) | 138 | 7 | 46 | 109
Vomiting (Gastrointestinal disorders) | 17 | 0 | 3 | 15
Upper respiratory tract infection (Infections and infestations) | 22 | 25 | 11 | 17
Urinary tract infection (Infections and infestations) | 13 | 21 | 9 | 6
Nasopharyngitis (Infections and infestations) | 14 | 6 | 4 | 4
Sinusitis (Infections and infestations) | 7 | 10 | 4 | 9
Injection site pain (General disorders) | 15 | 20 | 3 | 20
Injection site reaction (General disorders) | 18 | 3 | 2 | 14
Sunburn (Injury, poisoning and procedural complications) | 10 | 33 | 12 | 33
Abdominal pain upper (Gastrointestinal disorders) | 7 | 3 | 2 | 5
Diarrhea (Gastrointestinal disorders) | 7 | 3 | 4 | 7
Fatigue (General disorders) | 12 | 1 | 4 | 17
Injection site erythema (General disorders) | 8 | 1 | 2 | 2
Injection site pruritus (General disorders) | 7 | 1 | 2 | 4
Pain (General disorders) | 7 | 0 | 1 | 6
Dizziness (Nervous system disorders) | 10 | 1 | 0 | 10
Paresthesia (Nervous system disorders) | 7 | 0 | 0 | 4
Influenza (Infections and infestations) | 3 | 6 | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 5 | 4
Hot Flush (Vascular disorders) | 6 | 1 | 3 | 6
Somnolence (Nervous system disorders) | 1 | 1 | 1 | 6
Gastroenteritis Viral (Infections and infestations) | 4 | 7 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If there is no multi-site publication within 18 months after the Study has been completed or terminated at all Study sites, and all data have been received by Sponsor, the Site, and SMO shall have the right to publish its results from the Study for non-commercial purposes, if submitted to Sponsor for review 60 days prior to submission of publication. Publication must remove all confidential information and may be delayed by up to 180 days to allow Sponsor to protect its interests.